CLINICAL TRIAL: NCT06127836
Title: VISION (Vulvar ICG SLN Detection) Study: Near-Infrared Imaging With Indocyanine Green Injection for the Detection of Sentinel Lymph Nodes in Vulvar Cancer
Brief Title: Study of Near-Infrared Imaging With Indocyanine Green for Detection of Sentinel Lymph Nodes in People With Vulvar Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-310
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Vulvar Cancer
Keywords: Near-Infrared Imaging; Indocyanine Green; Sentinel Lymph Nodes; 23-310
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective study to evaluate the performance of near-infrared imaging with ICG injection, compared with lymphoscintigraphy, for the detection of the inguinofemoral SLN in patients with vulvar cancer.
Masking Description: Surgeons will be blinded to the results of the lymphoscintigraphy and will perform SLN biopsy in the operating room using near-infrared imaging with ICG injection. And the results will not be released until the consenting surgeon contacts the Nuclear Medicine team after attempting to identify the SLN by use of near-infrared imaging with ICG injection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients undergoing preoperative lymphoscintigraphy (Experimental): Patients will undergo radiocolloid lymphoscintigraphy before their surgery; the surgeon will be blinded to the results of this procedure. The surgeon will subsequently inject ICG in accordance with the SLN protocol in the operating room and will identify and remove the SLN by use of near-infrared imaging guidance only.
  Interventions: Procedure: ICG guided sentinel lymph node biopsy

INTERVENTIONS:
Procedure: ICG guided sentinel lymph node biopsy — The surgeon will subsequently inject ICG in accordance with the SLN protocol in the operating room and will identify and remove the SLN by use of near-infrared imaging guidance only. Once the surgeon has identified the SLN in this way, he or she will be unblinded to the results of the lymphoscintigraphy and will use the results of preoperative imaging and an intraoperative gamma counter to confirm the SLNs.

SUMMARY:
The purpose of this study is to compare two types of imaging for sentinel lymph node (SLN) mapping in people with early-stage vulvar cancer. The researchers will compare indocyanine green near-infrared (ICG-NIR) imaging with lymphoscintigraphy. All participants in this study will be scheduled for standard surgical treatment at Memorial Sloan Kettering Cancer Center (MSK). This surgical treatment includes SLN mapping (with both lymphoscintigraphy and ICG-NIR imaging) and SLN biopsy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Newly diagnosed with vulvar cancer and scheduled to undergo SLN biopsy (patients with squamous cell carcinomas and melanomas will be included)
* Primary tumor ≤4 cm in size
* For patients with squamous cell carcinoma, >1 mm of invasion is required

Exclusion Criteria:

* Clinically or radiographically enlarged inguinofemoral lymph nodes (if imaging is performed)
* Presence of distant metastases
* Absolute contraindication to radiocolloid Tc-99 or ICG
* Nonsquamous or nonmelanoma histologic subtype

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Vulvar cancer
Enrollment: 22 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
success of identifying the SLN | 18 months
  by use of near-infrared imaging with ICG injection. Patients will be eligible for assessment if they undergo attempted SLN mapping by lymphoscintigraphy and near-infrared imaging with ICG injection. The primary endpoint is the accurate identification of the SLN, defined as the uptake of ICG in the proximalmost draining lymph node in the inguinofemoral chain. Evaluate the ability of near-infrared imaging with ICG injection to detect the inguinofemoral SLN in patients with early-stage vulvar cancer, compared with radiocolloid lymphoscintigraphy, the current standard.

CONTACTS AND LOCATIONS:
Overall Officials: Vance Broach, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Houston Methodist Cancer Center (Data Collection Only), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm